CLINICAL TRIAL: NCT02934230
Title: The Prehabilitation Study: Exercise Before Surgery to Improve Patient Function in People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20160091
Record Dates: First submitted 2016-08-22; First posted 2016-10-14 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cancer; Frailty
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prehabilitation Group (Experimental): The intervention will be a home-based total-body exercise training program (prehabilitation) based on a protocol with proven efficacy in improving the function of non-frail surgical patients in less than 4 weeks of preoperative utilization.Prehabilitation will consist of 3 components: 1) strength training; 2) aerobic exercise and 3) flexibility. Prehabilitation will be prescribed as 1-hour sessions performed a minimum of 3 times per week. Intervention group patients will also be provided with nutritional advice. In addition to paper-based materials outlining the prehabilitation program, weekly prehabilitation teaching sessions will be held at our Cancer Centre for patients randomized to the intervention group, and activity logs and weekly phone calls will be used to measure compliance and to answer questions. During the final week of the program, patients will also participate in a brief qualitative interview over the phone to explore their experience with the program.
  Interventions: Behavioral: Prehabilitation Program
- Control Group (No Intervention): Patients randomized to the control group will be provided standard perioperative care as per our institutional standards. They will receive the World Health Organization (WHO) Global Recommendations for Physical Activity for Health for people 60 years and above pamphlet, as well as Canada's Food Guide. In-hospital perioperative care, and postoperative care, will be at the discretion of each patient's surgeon and anesthesiologist.

INTERVENTIONS:
Behavioral: Prehabilitation Program — Strength training: This component consists of 1 set of 10 repetitions of each exercise: a. push-ups (modified to the individual's level of function as either wall push-ups, knee push-ups, or full push-ups); b. seated row (performed with an elastic resistance band); c. chest fly (performed with an elastic resistance band); d. deltoid lift (performed with an elastic resistance band); e. biceps curls (performed with an elastic resistance band); f. triceps extensions (performed with an elastic resistance band); g. chair squats; h. hamstring curls; i. standing calf raises; j. abdominal crunches (modified to be performed seated in a chair)
  Aerobics: Walking for 20 minutes at moderate intensity.
  Flexibility: Chest, arm, leg and truck stretches, with each stretch to be held for 20 seconds, done for 2 repetitions.
  Arms: Prehabilitation Group

SUMMARY:
The rapid aging of the population means that anesthesiologists care for elderly patients with increasing regularity. Although age is an independent predictor for adverse postoperative outcomes, significant outcome variation exists among older surgical patients. Frailty, a syndrome that describes an aggregate susceptibility to adverse health outcomes due to age-, and disease-related deficits that accumulate across multiple domains is a key predictor of adverse postoperative outcomes in elderly patients. Frail surgical patients are at increased risk of complications, institutionalization, death, and are high healthcare resource users.

Multiple stakeholders, including anesthesiologists and patients, have identified improving the outcomes of older patients and preoperative exercise training (prehabilitation) as 2 of the 10 most important areas for future perioperative research. Physical vulnerability is an important aspect of the frailty syndrome, and may be amenable to structured exercise therapy. However, the evidence for preoperative exercise training (prehabilitation) improving postoperative outcomes is obscured by methodological limitations and a focus on non-elderly patients. Recently, evidence has emerged that older and sicker patients may benefit most from prehab, however, this hypothesis has not been formally tested.

Because the complex needs of frail perioperative patients require a longitudinal and multidisciplinary approach, the investigators are developing a perioperative surgical home for the frail elderly (PSH-Frail). Development of the PSH-Frail is supported by a robust data collection system, including linkage of prospectively collected data to health administrative data infrastructure to improve efficiency and long-term follow up.

The investigators hypothesize that prehabilitation will be a vital intervention supported by the PSH frail, however, high quality evidence from randomized trials is needed to support its efficacy. Therefore, the investigators propose a single center randomized controlled trial of prehabilitation of frail elderly patients having elective abdominal and thoracic cancer surgery to improve postoperative function (primary outcome), and to decrease postoperative resource utilization (secondary outcomes).

DETAILED DESCRIPTION:
Frailty is a key risk factor for adverse outcomes among the increasingly large number of older patients presenting for surgery. The complexity and risk profile of frail patients makes them a population who may derive significant benefit from the multidisciplinary and continuous care provided by a Perioperative Surgical Home (PSH) model of care. Development of an evidence-based PSH for the frail elderly (PSH-Frail) is the overarching goal of the investigator's research program. However, the PSH-Frail is a complex intervention, and will require high quality evidence to support inclusion of specific processes and interventions into the overall framework.

To date, the investigator's research group has undertaken prospective studies to support the routine and accurate identification of frail patients before surgery. The next step in the development of the PSH-Frail is testing interventions to improve the outcomes of frail elderly surgical patients. The role of preoperative exercise training (prehabilitation) in improving postoperative outcomes is a priority research area in perioperative medicine, and may provide its most significant impact in frail elderly patients. However, this hypothesis has not been formally tested.

Study design:

A single center, parallel arm randomized controlled trial of home-based prehabilitation vs. standard perioperative care in frail elderly patients undergoing elective surgery for intraabdominal cancer will be conducted. This will be a superiority trial to test the hypothesis that home-based prehabilitation will result in improved postoperative functional outcomes compared to standard care. This protocol is described in keeping with the Standard Protocol Items: Recommendations for Intervention Trials (SPIRIT) guidelines).

Study setting:

This study will be performed at The Ottawa Hospital (TOH), a 900-bed tertiary care academic health sciences center serving a catchment area of 1.2 million people. TOH is the regional cancer referral center for the Eastern portion of the Canadian province of Ontario. On average, cancer patients are seen 4 weeks prior to surgery (as this is a provincial benchmark for cancer care).

Sample size:

To detect a clinically important 25 meter difference in the primary outcome between study arms, using a two-sided test at the 5% level of significance with 80% power, and assuming a standard deviation of 55 meters based on a previously published trial, we will require 77 patients per arm. To account for up to 20% attrition we will enroll 100 patients per arm.

Recruitment:

Patients will be recruited from the investigator's hospital's Cancer Assessment Center. Following cancer diagnosis, patients are seen by a surgeon 4 weeks prior to their scheduled operation. Following surgical assessment and confirmation of the decision to operate, patients who consent to consideration for research contact, and who meet all inclusion criteria except for frailty score, will be assessed by a trained clinician or clinical assistant using the Clinical Frailty Scale (CFS). Patients who score >4/9 on the CFS will then be randomized after providing written informed consent.

Intervention:

The intervention will be a home-based total-body exercise training program (henceforth referred to as prehabilitation) based on a protocol with proven efficacy in improving the function of non-frail surgical patients in less than 4 weeks of preoperative utilization. Prehabilitation will consist of 3 components: 1) strength training; 2) aerobic exercise and 3) flexibility. Prehabilitation will be prescribed as 1-hour sessions performed a minimum of 3 times per week.

Control:

Patients randomized to the control group will be provided standard perioperative care as per institutional standards. Patients will receive the World Health Organization (WHO) Global Recommendations for Physical Activity for Health for people 65 years and above pamphlet, as well as Canada's Food Guide. In-hospital perioperative care, and postoperative care, will be at the discretion of each patient's surgeon and anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* scheduled to undergo elective surgery for intraabdominal or thoracic cancer
* diagnosed with frailty based on the Clinical Frailty Scale (CFS; score of >4/9 defines frailty)

Exclusion Criteria:

* cannot communicate in written or oral form in official languages serviced by TOH (English or French)
* unwilling to participate in home-based prehabilitation
* major cardiac risk factors
* scheduled to undergo surgery in fewer than 3 weeks from randomization

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative functional capacity | 30 days after surgery
  Functional capacity at baseline (surgical assessment typically 4 weeks prior to surgery) compared to postoperative functional capacity 30 days after surgery. The primary outcome of this study will be postoperative functional capacity, specifically the 6-minute walk test 30 days after surgery. A clinically relevant difference in this outcome is a change of 25 meters walked over 6 minutes.

SECONDARY OUTCOMES:
Functional Mobility | 30 days after surgery
  Functional outcomes will be assessed using the Short Physical Performance Battery (SPPB).This is a validated, objective assessment, developed by National Institute on Ageing, to evaluate lower extremity functioning in older individuals through assessment of balance, gait speed and lower limb functional strength; each domain is assessed on a 4-point scale, and the overall performance is rated on a cumulative 12-point scale. Participants will complete this at baseline (surgical assessment typically 4 weeks prior to surgery) and at their post-operative surgical follow-up (approximately 30 days after surgery).
Patient-reported health outcomes and adverse events: Health Related Quality of Life - health state | 30 and 90 days after surgery
  Measured using the EQ-5D30 (5-level version). The EQ-5D assesses domains of self-perceived mobility, self-care, usual activity participation, pain/discomfort, and anxiety depression which is captured as a overall health state score.
Patient-reported health outcomes and adverse events: Health Related Quality of Life | 30 and 90 days after surgery
  Measured using the EQ-5D30 (5-level version). The EQ-5D also uses a self-report 0-100 point scale relating the person's current health status to their best imaginable status
Patient-reported health outcomes and adverse events: Disability Free Survival | 30 and 90 days after surgery
  Measured using the WHODAS 2.0 instrument, a 30-day look-back multidimensional disability scale that is validated in a variety of disease states, including postoperatively.
Patient-reported health outcomes and adverse events: Adverse Events | Within 365 days after surgery
  Based on the National Surgical Quality Improvement Program definitions for medical complications, the type of medical complication will be collected.
Patient-reported health outcomes and adverse events: Adverse Events | Within 365 days after surgery
  Based on the National Surgical Quality Improvement Program definitions for surgical complications, the type of surgical complication will be collected.
Patient-reported health outcomes and adverse events: Adverse Events | Within 365 days after surgery
  The number of participants who experience all-cause mortality will be collected.
Healthcare resource utilization: hospital length of stay | Within 365 days after surgery
  Number of days in hospital post-operatively
Healthcare resource utilization: proportion of patients discharged to an institution, readmissions within 30 days of discharge | Within 365 days after surgery
  Number of patients discharged to an institution and/or re-admitted post-operatively
Healthcare resource utilization: total healthcare costs | Within 365 days after surgery
  Amount of healthcare dollars spent will be generated using a validated algorithm in our administrative data

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I McIsaac, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McIsaac DI, Neilipovitz N, Bryson GL, Gagne S, Huang A, Lalu M, Lavallee LT, Moloo H, Power B, Scheede-Bergdahl C, van Walraven C, McCartney CJL, Taljaard M, Hladkowicz E. Home-based exercise prehabilitation to improve disease-free survival and return to intended oncologic treatment after cancer surgery in older adults with frailty: a secondary analysis of a randomized trial. Can J Anaesth. 2024 Nov;71(11):1525-1534. doi: 10.1007/s12630-024-02835-w. Epub 2024 Sep 5. PMID 39237725
- [Derived] McIsaac DI, Hladkowicz E, Bryson GL, Forster AJ, Gagne S, Huang A, Lalu M, Lavallee LT, Moloo H, Nantel J, Power B, Scheede-Bergdahl C, van Walraven C, McCartney CJL, Taljaard M. Home-based prehabilitation with exercise to improve postoperative recovery for older adults with frailty having cancer surgery: the PREHAB randomised clinical trial. Br J Anaesth. 2022 Jul;129(1):41-48. doi: 10.1016/j.bja.2022.04.006. Epub 2022 May 17. PMID 35589429
- [Derived] McIsaac DI, Saunders C, Hladkowicz E, Bryson GL, Forster AJ, Gagne S, Huang A, Lalu M, Lavallee LT, Moloo H, Nantel J, Power B, Scheede-Bergdahl C, Taljaard M, van Walraven C, McCartney CJL. PREHAB study: a protocol for a prospective randomised clinical trial of exercise therapy for people living with frailty having cancer surgery. BMJ Open. 2018 Jun 22;8(6):e022057. doi: 10.1136/bmjopen-2018-022057. PMID 29934394